CLINICAL TRIAL: NCT03476083
Title: Tenofovir Disoproxil Fumarate in Combination of Hepatitis B Vaccine With the Omission of Immune Globulin to Prevent Hepatitis B Transmission in Mother With High Viral Load: A Multi-Center, Prospective, Randomized and Open-Label Study
Brief Title: Tenofovir Disoproxil Fumarate in Combination of Hepatitis B Vaccine for Preventing Hepatitis B Vertical Transmission
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New Discovery LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: US-G10-P616; (2018) 462 No: HGRSL20180412 (Other: Ministry of Science and Technology of China, HGRM Office)
Record Dates: First submitted 2018-03-18; First posted 2018-03-23 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis B Infection; Congenital Malformation; Birth Defect; Viremia; Chronic Infection
Keywords: Mother to Child Transmission; Hepatitis B Infection; Congenital Defects or Malformation; Hepatitis B Vaccine; Hepatitis B Immunoglobulin; Pregnancy; Antiviral Treatment
MeSH Terms: conditions — Hepatitis B; Congenital Abnormalities; Viremia; Persistent Infection | interventions — Tenofovir; hepatitis B hyperimmune globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): This is the experimental group. Participating mothers will receive Tenofovir Disoproxil Fumarate (TDF) 300 mg oral daily, starting at gestational weeks 14-16 and continue until delivery. The mothers will be followed together with their infants until postpartum week 28. Infants will receive hepatitis B vaccine at birth and additional hepatitis B (HBV) vaccine at the age of week 4 and week 24. HBIg will be omitted for the infants in this group.
  Interventions: Drug: Tenofovir Disoproxil Fumarate (TDF) 300 mg oral daily.
- Group B (Active Comparator): This is the comparative group. Participating mothers will receive Tenofovir Disoproxil Fumarate (TDF) 300 mg oral daily, starting at gestational weeks 28 and continue until delivery. Patients in group B will have similar follow-up schedules as those in the experimental group. Infants will receive hepatitis B vaccine plus HBIg at birth and additional hepatitis B vaccine at the age of week 4 and week 24.
  Interventions: Drug: Tenofovir Disoproxil Fumarate (TDF) 300 mg oral daily.

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate (TDF) 300 mg oral daily. — All mothers will receive TDF therapy. However, group A will initiate TDF at the gestational week of 14-16, while group B will initiate TDF at the gestational week of 28. All infants will receive a series of three hepatitis B vaccines (at birth, age of weeks 4 and 24). In addition, the infants in the group B will receive HBIg injection at birth.
  Other Names: HBIg 200 IU im for infants in the group B; HBV vaccine 10 ug im for all infants

SUMMARY:
Immunoprophylaxis with two hepatitis B vaccinations following the hepatitis B immune globulin (HBIg) and hepatitis B vaccine at birth is largely effective in protecting infants from hepatitis B virus (HBV) infection. However, hepatitis B infection due to immunoprophylaxis failure often occurs in approximately 10% of infants who are born to highly viremic mothers with HBeAg-positive. Maternal HBV DNA > 200,000 IU/mL is the major independent risk for mother-to-child transmission (MTCT). A recent randomized controlled trial has shown that Tenofovir Disoproxil Fumarate (TDF) use during the third trimester of pregnancy could safely reduce the rate of MTCT with few adverse effects when combined with the administration of the standard immunoprophylaxis to the infants. However, HBIg is expensive and not available in many developing countries, resulting approximately 30% of infant infection when they received only HBV vaccination. The present study aims to investigate if highly viremic mothers who are treated with TDF from the second trimester to delivery in combination of infant's standard series of HBV vaccinations (omission of HBIg) have a comparable MTCT rates, when compared to those of mothers who receive TDF at the third trimester in combination of infant's standard HBV vaccinations and a birth dose of HBIg.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, open-label and parallel two arm study starting from week 14-16 of pregnancy to post-partum week 28. The enrollment from approximately 7 centers will be in blocks for sample balance. By using the randomized table, 280 HBeAg-positive pregnant women with chronic hepatitis B (CHB) will be randomized in a 1:1 ratio in to two arms. Group assignments will be also stratified by the maternal HBV DNA levels >9 log10 versus ≤ 9 log10 IU/mL.

Group A: This is the experimental group. Participating mothers will receive TDF (oral 300 mg tablet daily) starting at gestational weeks 14-16 and continue until delivery. The mothers will be followed together with their infants until postpartum week 28. Infants will receive hepatitis B vaccine at birth (within 12 hours) and additional hepatitis B vaccine at the age of week 4 and week 24. HBIg will be omitted for the infants in this group. However, the birth dose of HBIg will be provided to infants born to mothers who have poor control of maternal viremia (i.e. the levels of HBV DNA >200,000 IU/mL before delivery). Group B: This is the comparative group. Participating mothers will receive TDF (oral 300 mg tablet daily) starting at gestational weeks 28 and continue until delivery. Patients in group B will have similar follow-up schedules as those in the experimental group. Infants will receive hepatitis B vaccine plus HBIg at birth (within 12 hours) and additional hepatitis B vaccine at the age of week 4 and week 24.

ELIGIBILITY:
Inclusion Criteria:

* HBeAg-positive CHB mothers
* Age of 20-35 years old
* Serum HBV DNA levels > 200,000 IU/mL
* Gestational age between 12-14 weeks.
* Both mother and father of the child have the ability to understand and are willing to consent to the study.

Exclusion Criteria:

* Co-infection with (HIV)-1, or hepatitis A, C, D, E or sexual transmitted diseases (STD)
* History of abortion or congenital malformation in a prior pregnancy
* Treatment experience (except when antivirals were used for MTCT prevention in a previous pregnancy and discontinued >6 months prior to the current pregnancy)
* History of renal dysfunction; evidence of liver cancer or decompensation
* Estimated creatinine clearance (CLCr) <100 mL/min (using the Cockcroft-Gault method based on serum creatinine and ideal body weight)
* Hypo-phosphoremia; hemoglobin <8 g/dL; neutrophil count <1,000//μL; alanine aminotransferase >5 times upper limit of the normal; total bilirubin >2 mg/dL; albumin <25gm/L;
* Clinical signs of threatened miscarriage
* Ultrasonographic evidence of fetal deformity
* Concurrent treatment with nephrotoxic drugs, steroids, cytotoxic drugs, nonsteroidal anti-inflammatory drugs, or immune modulators;
* Recipient of solid organ or bone marrow transplant
* Significant renal, cardiovascular, pulmonary, neurological disease or other health conditions in the opinion of the investigator
* Fetus's biological father had CHB infection

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 280 (Estimated)
Dates: Start 2018-06-10 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Assessment on the proportion of infants who are infected with hepatitis B at the age of 28 weeks in the two groups | From the date of birth to age of 28 weeks.
  Compare MTCT rates between the two study groups and demonstrate non-inferiority in efficacy. MTCT rate is defined as the proportion of infants with serum HBV DNA >20 IU/mL and/or HBsAg positivity at 28 weeks of age.

SECONDARY OUTCOMES:
Assessment on congenital defects and/or malformation rates in each infant group for comparison | From the date of birth to age of 28 weeks.
  Congenital defects and/or malformation rates are defined as the proportion of infants with the aforementioned abnormalities discovered during the study period.
Assessment on the reduction of maternal HBV DNA levels at delivery | From the date of randomization until delivery.
  Assess the reduction of maternal HBV DNA levels at delivery when compared to the baseline before initiating TDF.
Maternal serological outcomes during the study: Percentage of mothers who loss/seroconversion of HBsAg or/and HBeAg during the study | From the date of randomization until postpartum week 28.
  Assess the percentage of mothers who loss/seroconversion of HBsAg or/and HBeAg during the study.
Adverse events of both mothers and infants | From the date of screening until postpartum week 28.
  Assess the percentage of mothers or infants who have adverse events during the study.
Tolerability of TDF therapy: Percentage of mothers who discontinue on TDF therapy due to the adverse event(s) during the study | From the date of randomization until delivery.
  Assess the percentage of mothers who discontinue on TDF therapy due to the adverse event(s) during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Q Pan, MD, Study Chair — Leading Principle Investigator, NYU Langone Health, NYU School of Medicine, NY; Erhei Dai, MD, Study Director — The Fifth Hospital of Shijiazhuang, Shijiazhuang, Hebei Province, China
Locations (7):
- China (7):
  - Beijing Youan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Guangzhou Women and Children's Medical Center, Guangzhou Medical University, Guangzhou, Guangdong
  - The Fifth Hospital of Shijiazhuang, Shijiazhuang, Hebei
  - Shijiazhuang Maternal and Child Health Care Hospital, Shijiazhuang, Hebei
  - Department of Infectious Diseases, the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The Third People's Hospital of Shenzhen, Shenzhen, Shenzhen

REFERENCES:
- [Background] Ott JJ, Stevens GA, Wiersma ST. The risk of perinatal hepatitis B virus transmission: hepatitis B e antigen (HBeAg) prevalence estimates for all world regions. BMC Infect Dis. 2012 Jun 9;12:131. doi: 10.1186/1471-2334-12-131. PMID 22682147
- [Background] Pan CQ, Duan ZP, Bhamidimarri KR, Zou HB, Liang XF, Li J, Tong MJ. An algorithm for risk assessment and intervention of mother to child transmission of hepatitis B virus. Clin Gastroenterol Hepatol. 2012 May;10(5):452-9. doi: 10.1016/j.cgh.2011.10.041. Epub 2011 Nov 9. PMID 22079509
- [Background] Pande C, Sarin SK, Patra S, Kumar A, Mishra S, Srivastava S, Bhutia K, Gupta E, Mukhopadhyay CK, Dutta AK, Trivedi SS. Hepatitis B vaccination with or without hepatitis B immunoglobulin at birth to babies born of HBsAg-positive mothers prevents overt HBV transmission but may not prevent occult HBV infection in babies: a randomized controlled trial. J Viral Hepat. 2013 Nov;20(11):801-10. doi: 10.1111/jvh.12102. Epub 2013 Apr 23. PMID 24168259
- [Background] Lee LY, Aw MM, Saw S, Rauff M, Tong PY, Lee GH. Limited benefit of hepatitis B immunoglobulin prophylaxis in children of hepatitis B e antigen-negative mothers. Singapore Med J. 2016 Oct;57(10):566-569. doi: 10.11622/smedj.2015194. Epub 2015 Dec 29. PMID 26778725
- [Background] Machaira M, Papaevangelou V, Vouloumanou EK, Tansarli GS, Falagas ME. Hepatitis B vaccine alone or with hepatitis B immunoglobulin in neonates of HBsAg+/HBeAg- mothers: a systematic review and meta-analysis. J Antimicrob Chemother. 2015 Feb;70(2):396-404. doi: 10.1093/jac/dku404. Epub 2014 Oct 31. PMID 25362571
- [Background] Pan CQ, Duan Z, Dai E, Zhang S, Han G, Wang Y, Zhang H, Zou H, Zhu B, Zhao W, Jiang H; China Study Group for the Mother-to-Child Transmission of Hepatitis B. Tenofovir to Prevent Hepatitis B Transmission in Mothers with High Viral Load. N Engl J Med. 2016 Jun 16;374(24):2324-34. doi: 10.1056/NEJMoa1508660. PMID 27305192
- [Background] Pan, C. Q.; Chang, T. T.; Bae, S. H.; Brunetto, M.; Coffin, C.; Lau, A.; Mo, S.; Flaherty, J. F.; Gaggar, A.; Subramanian, G. M.; Nguyen, M. H.; Gurel, S.; Thompson, A.; Gane, E. J. Viral kinetics in women of child bearing potential with chronic hepatitis B virus following treatment with tenofovir alafenamide or tenofovir disoproxil fumarate. J Hepatol. 2017;66 S258-S259.
- [Derived] Pan CQ, Dai E, Mo Z, Zhang H, Zheng TQ, Wang Y, Liu Y, Chen T, Li S, Yang C, Wu J, Chen X, Zou H, Mei S, Zhu L. Tenofovir and Hepatitis B Virus Transmission During Pregnancy: A Randomized Clinical Trial. JAMA. 2025 Feb 4;333(5):390-399. doi: 10.1001/jama.2024.22952. PMID 39540799